CLINICAL TRIAL: NCT05310695
Title: A Naturalistic Efficacy Trial of the Norwegian Sickness Absence Clinic for Patients With Common Mental Disorder and Musculoskeletal Disorders
Brief Title: A Naturalistic Trial of the Norwegian Sickness Absence Clinic. The NSAC Efficacy Study
Acronym: NSAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: University Hospital of North Norway (Other); Helsepartner Rehabilitering AS (Alta, Norway) (Unknown); Helgeland Hospital Trust (Other); Finnmarkssykehuset HF (Kirkenes, Norway) (Unknown); UiT The Arctic University of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/1168-XX
Record Dates: First submitted 2022-03-16; First posted 2022-04-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Musculoskeletal Disorder; Anxiety Disorders; Depression; Fatigue; Pain; Occupational Exposure; Work Related Stress; Workplace Bullying; Employment; Sickness Absence; Return to Work
Keywords: Return to work; Sickness absence; Nudge; Barriers for return to work; Motivation for work; Demand and control; Work/family conflict; Bullying
MeSH Terms: conditions — Musculoskeletal Diseases; Anxiety Disorders; Depression; Fatigue; Pain; Occupational Stress; Bullying

STUDY DESIGN:
Intervention Model Description: Patients are randomized to either of three intervention arms:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NSAC rapid: treatment at the NSAC at- or within 4 weeks (Active Comparator): NSAC service delivered according to ordinary procedures, 4 weeks after referral.
  Interventions: Other: NSAC - rapid
- NSAC ordinary: treatment at the NSAC after 10-14 weeks (Active Comparator): NSAC service delivered according to ordinary procedures, 10-14 weeks after referral, by and large equivalent to current waiting time
  Interventions: Other: NSAC - ordinary
- NSAC - active control (Active Comparator): Monodisciplinary examination at the NSAC close to diagnosis-specific deadline for examination as suggested by guidelines (8-26 weeks, the majority at the end of this interval)
  Interventions: Other: NSAC - active control

INTERVENTIONS:
Other: NSAC - rapid — NSAC is an outpatient service delivered under the auspices of the specialist health care sector to patients currently on sick leave or at risk for long-term sickness absence. The service is staffed by medical doctors specialising in muskuloskeletal health, physiotherapists, psychologists and welfare sector counsellors, and aims to provide patients with a multi-diciplinary clarification or treatment of problems with the intent of improved function and return to work. Clinicians are provided survey information on the patients potential health problems, motivation for work, barriers for return to work and work environment prior to consultation. In this intervention arm, patients are offered treatment within 4 weeks of referral.
  Arms: NSAC rapid: treatment at the NSAC at- or within 4 weeks
Other: NSAC - ordinary — NSAC is an outpatient service delivered under the auspices of the specialist health care sector to patients currently on sick leave or at risk for long-term sickness absence. The service is staffed by medical doctors specialising in muskuloskeletal health, physiotherapists, psychologists and welfare sector counsellors, and aims to provide patients with a multi-diciplinary clarification or treatment of problems with the intent of improved function and return to work. Clinicians are provided survey information on the patients potential health problems, motivation for work, barriers for return to work and work environment prior to consultation. In this intervention arm, patients are offered treatment at 10-14 weeks after referral.
  Arms: NSAC ordinary: treatment at the NSAC after 10-14 weeks
Other: NSAC - active control — The active control intervention is provided by the NSAC personnel, but patients are offered a single monodisciplinary examination close to the end of the diagnosis-specific deadline suggested in guidelines, which will vary between 8-26 weeks. Employment counsellors may not be involved in consultations, other cross-disciplinary consultations are restricted, and work-related factors are not to be focused on during examination. Clinicians are provided survey information only on the patient's potential health problems prior to consultation. Patients are provided a health-focused examination, with the aim of symptom-relief.
  Arms: NSAC - active control

SUMMARY:
The Norwegian Sickness Absence Clinic (NSAC) is a publicly funded specialist outpatient health service, which is uniquely available for the work force. The overall aim of the NSAC is prevention of sickness absence, promote return to work (RTW) among those on sickness absence and prevent long term disability benefit dependency. In addition to being a health service, the NSAC has a focus on work and functional recovery, including also non-health related factors. Patients can be referred by general practitioners for mental health problems and musculoskeletal problems. The NSAC has a lower threshold for severity than specialist health services generally, and in particular for mental health problems. The efficacy of this service is unknown.

The NSAC Efficacy Study is a randomized controlled multicentre trial which aims to assess the effect of the NSAC service. "Helse i Arbeid" is the Norwegian name for NSAC, and the Norwegian abbreviation is "HiA". The Norwegian study name is HIANOR.

The NSAC Efficacy Study involves five different NSACs across northern Norway, and will recruit 2500 patients, randomized to in equal proportions to three treatment arms:

1. NSAC - rapid: treatment at the NSAC at- or within 4 weeks
2. NSAC - ordinary: treatment at the NSAC after 10-14 weeks
3. NSAC - active control: monodisciplinary examination at the NSAC close to diagnosis-specific deadline for examination as suggested by guidelines (8-26 weeks, the majority at the end of this interval) The overall aim is to assess the effect of the NSAC service, with the hypothesis that the NSAC service is superior to what resembles treatment as usual (TAU) for outcomes such as return to work or improved health (waiting list control). Many of the diagnoses or problems for which patients are referred to the NSACs naturally improve regardless of health interventions, and - as of date - no research has been conducted to assess the efficacy of the service.

DETAILED DESCRIPTION:
The Norwegian Sickness Absence Clinic (NSAC) is a publicly funded specialist outpatient health service, which is uniquely available for the work force. The overall aim of the NSAC is prevention of sickness absence, promote return to work (RTW) among those on sickness absence and prevent long term disability benefit dependency. In addition to being a health service, the NSAC has a focus on work and functional recovery, including also non-health related factors. Patients can be referred by general practitioners for mental health problems and musculoskeletal problems. The NSAC has a lower threshold for severity than specialist health services generally, and in particular for mental health problems. The efficacy of this service is unknown.

The NSAC Efficacy Study is part of a broader project, the Norwegian Sickness Absence Clinic Study (NSACS). The NSACS currently has two sources of funding: Northern Norway Regional Health Authority and The Norwegian Labour and Welfare Administration and involves two RCTs: NSAC Efficacy and NSAC Nudge and fifteen work packages concerning health economics, scalability, implementation, profiling of patient groups, and non-RCT related research questions to improve understanding of the patient group and their challenges. To do this the project will use patient survey data, clinician-reported procedures, opinions and outcomes, linked to registry data for work benefits and health service use. The randomized controlled trial NSAC Efficacy is the subject of this trial registration.

The NSAC Efficacy Study is a naturalistic randomized controlled multicentre trial, carried out in northern Norway and involving five NSACs. The study invites 2500 patients, randomized to either of three treatment arms:

1. NSAC rapid: treatment at the NSAC at- or within 4 weeks
2. NSAC ordinary: treatment at the NSAC after 10-14 weeks
3. NSAC - active control: monodisciplinary examination at the NSAC close to diagnosis-specific deadline for examination as suggested by guidelines (8-26 weeks, the majority at the end of this interval)

The NSACs are staffed by teams of medical doctors specializing in physical medicine and rehabilitation, psychologists, physiotherapists, and employment counsellors with experience from case management in the Norwegian Labor and Welfare Administration (NAV).

All patients are asked to complete an electronic survey about their mental health and musculoskeletal pain, work conditions, motivation for work and barriers for return to work (RTW). The control group only completes the survey on health, and only on either mental health or musculoskeletal pain, according to referral diagnosis.

The survey tool manages the randomization algorithm.

The NSAC is a relatively new clinical service, available for the labour force, and publicly funded with the intention to reduce sickness absence and prevent retirement from the labour force and transitions to disability benefits. The NSAC clinic welcomes patients with the most common diagnoses for sickness absence and is supposed to have a low threshold.

There is no single alternative clinical service for similar patients outside the labour force, thus no single treatment as usual (TAU) alternative. Service availability will depend on diagnosis and severity:

* The majority of patients eligible for treatment in the NSAC referred with mental disorders would not be eligible for treatment in specialist psychiatric services as conditions in most cases would be too mild. The most common treatment alternative would be treatment at the general practitioners.
* For patients referred for musculoskeletal problems, some may be eligible for consultations and treatment at physical medicine and rehabilitation outpatient clinics. For those not eligible, the general practitioner is the most common alternative, and other options such as private physiotherapists. Eligibility criteria may vary between catchment areas.
* All alternatives to the NSAC would be without employment counsellors, little cross disciplinary assessment, and little to no focus on work and functional rehabilitation.

The active control group aims to be comparable to TAU, and differs from the NSAC in the following respects:

1. Patients receive a monodisciplinary examination from either a doctor, physiotherapist of psychologist at the NSAC. The focus of the examination is on health-related factors. The patients will not receive further follow-up at the clinic beyond the first examination. Upon indication, the patient is referred to other treatment or examination outside of the NSAC.
2. Employment counsellors are not involved in patient consultations or in discussions about patients.
3. Patients in the active control group will not be posed questions concerning work, motivation for work or barriers for return to work. Patients will during registration in Tivian be classified as having predominantly either musculoskeletal- or common mental disorders, and this will dictate the type of questions posed: musculoskeletal patients will be asked questions on musculoskeletal factors but not psychological factors, while patients will common mental disorders will be asked questions about psychological factors but not musculoskeletal issues. For patients being examined by a psychologist, if issues concerning musculoskeletal health arise, the patient is asked to discuss these with his/her GP. If issues concerning mental health arise which requires competence beyond what the physiotherapist possesses, the physiotherapist may confer with the medical doctor at NSAC.
4. The clinician is not to take initiative to discussing work-related factors with the patient, and as far as possible avoid these becoming central topics of the consultation. If the patient on his/her own initiative brings up such topics, the clinician is not restricted from addressing them.
5. Employment counsellors are not part of patient discussions prior to examination.
6. Meetings or discussions about patients are kept within profession; i.e. a physiotherapist is allowed to discuss his/her patient with other physiotherapists if need be.

The data necessary to answer the research questions are gathered from national registries via personal identifier, registry data on population level, questionnaires filled out by the patient (data on health and working conditions) and questionnaires filled out by the clinician (data on number of treatments, diagnosis, professions involved, and types of treatment provided).

The patient questionnaire covers 9 themes, split in two sections. Section 1 covers health, and includes musculoskeletal problems, mental health, and other health related issues (such as alcohol consumption, medication, and physical activity). Section 2 includes working conditions (including inter alia questions on social support, work/family conflict and bullying), barriers for RTW, labour market affiliation, other personal aspects (such as demography and motivation for work), questionnaires for health economic evaluation (such as the EQ-5D) and expectations for treatment.

By and large the questionnaire consists of test batteries which have been validated for specific topics. To reduce the number of questions posed to each patient, the baseline questionnaire will employ index questions which have proven psychometric properties in terms of factor loading or similar, meaning that if a problem on a specific topic such as neck pain is not indicated, the patient will not be presented with the Neck Disability Index questionnaire. The patient questionnaires will be filled out electronically at before first treatment and at 6- and 12 months after first treatment. In addition, before treatments, patients will be given shorter versions of the same questionnaire to be filled out at the clinic. These shorter questionnaires will consist of questions to which the patient at baseline indicated a high score, and thus includes more relevant information to the clinician.

In the NSAC Efficacy Study, receiving treatment at NSACs presupposes consent to participate in research, as the effect of the treatment is as of date unknown. Hence, receiving treatment at the NSAC is not necessarily superior to other available health services. Other available health services that may be utilized by patients serving in the control groups include mono-disciplinary treatment by physiotherapists, psychologists, general practitioners, gyms, electronically delivered self-help tools etc. All patients referred to NSACs will be offered treatment, but patients that decline to participate in research are provided an examination in line with randomization arm #3.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be considered eligible for treatment at the NSAC by the admission team at the NSAC.

Exclusion Criteria:

* Patients considered too healthy for treatment at the NSAC, i.e. not within target group
* Patients considered too sick for treatment at the NSAC, i.e. not within target group
* Patients that do not have a diagnosis that is relevant for treatment at the NSAC, i.e. not within target group
* Patients otherwise considered not within target group for the measure
* Patients which were included in the NSAC Nudge trial (clinicaltrials identifier: NCT05006976)
* Patients which are secondary referred from other departments/clinics within the hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2034-10 (Estimated)

PRIMARY OUTCOMES:
Functional recovery: employment | 12 months post baseline survey
  Employment during first 365 days post baseline survey, based on registry data and self-report.
Functional recovery: sickness absence | 12 months post baseline survey
  Sickness absence during first 365 days post baseline survey, based on registry data and self-report.
Functional recovery: application for rehabilitation benefits | 12 months post baseline survey
  Application for rehabilitation benefits during first 365 days post baseline survey, based on registry data and self-report.
Functional recovery: employment long term | 5 and 10 years post baseline survey
  Employment during 5-and 10-year period post baseline survey, all based on registry data.
Functional recovery: sickness absence long term | 5 and 10 years post baseline survey
  Sickness absence during 5-and 10-year period post baseline survey, all based on registry data.
Functional recovery: rehabilitation benefits long term | 5 and 10 years post baseline survey
  Rehabilitation benefits during 5-and 10-year period post baseline survey, all based on registry data.
Functional recovery: disability benefits long term | 5 and 10 years post baseline survey
  Disability benefits during 5-and 10-year period post baseline survey, all based on registry data.

SECONDARY OUTCOMES:
Mental health | 12 months post baseline survey
  Changes in self-reported mental health between baseline survey and 6- and 12 months post baseline survey, measured using the Hopkins Symptoms Checklist - 10 (HSCL-10).
Anxiety | 12 months post baseline survey
  Changes in self-reported anxiety between baseline survey and 6- and 12 months post baseline survey, measured using the Beck Anxiety Inventory (BAI). The instrument is provided to patients upon indication, defined as a HSCL-10 score > 1.4
Depressive symptoms | 12 months post baseline survey
  Changes in self-reported depression between baseline survey and 6- and 12 months post baseline survey, measured using the Beck Depression Inventory (BDI). The instrument is provided to patients upon indication, defined as a HSCL-10 score > 1.4
Sleep | 12 months post baseline survey
  Changes in self-reported sleep between baseline survey and 6- and 12 months post baseline survey, measured using 3 questions commonly used to diagnose sleeping disorder according to the DSM-IV criteria for insomnia.
Health Anxiety | 12 months post baseline survey
  Changes in self-reported health anxiety between baseline survey and 6- and 12 months post baseline survey, measured using the Whitely Index. All patients are asked the first question in the test battery, and the entire instrument is provided to patients with a score of >3 on this question
Subjective health complaints | 12 months post baseline survey
  Changes in subjective healthbetween baseline survey and 6- and 12 months post baseline survey, measured using a modified version of the Ursin Health Inventory.
Back pain | 12 months post baseline survey
  Changes in self-reported back pain between baseline survey and 6- and 12 months post baseline survey, measured using the Oswestry Disability Index (ODI). All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided questions on localization of pain. In case of back pain, patients are provided the ODI.
Neck pain | 12 months post baseline survey
  Changes in self-reported neck pain between baseline survey and 6- and 12 months post baseline survey, measured using the Neck Disability Index (NDI). All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided questions on localization of pain. In case of neck pain, patients are provided the NDI.
Pain intensity | 12 months post baseline survey
  Changes in self-reported pain intensity between baseline survey and 6- and 12 months post baseline survey, measured using a visual analogue scale scored between 0 and 10. All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided questions on pain intensity during rest and activity.
Fear avoidance | 12 months post baseline survey
  Changes in self-reported fear avoidance between baseline survey and 6- and 12 months post baseline survey, measured using the Fear Avoidance Beliefs Questionnaire (FABQ). All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided the FABQ.
Physical activity | 12 months post baseline survey
  Changes in self-reported level of physical between baseline survey and 6- and 12 months post baseline survey, measured using the Saltin-Grimby Physical Activity Level Scale (SGPALS).
Fatigue | 12 months post baseline survey
  Changes in self-reported fatigue between baseline survey and 6- and 12 months post baseline survey, measured using the Fatigue Assessment Scale. All patients are asked the first question in the test battery, and the entire instrument is provided to patients with a score of ≥ 3 on this question
Pain localization | 12 months post baseline survey
  Changes in self-reported localization of pain between baseline survey and 6- and 12 months post baseline survey. All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided questions on localization of pain.
Cause of pain | 12 months post baseline survey
  Changes in self-reported cause of pain between baseline survey and 6- and 12 months post baseline survey. All patients are asked whether they suffer from musculoskeletal pain, and if present, they are provided questions on the believed cause of pain.
Self-reported diagnosis | 12 months post baseline survey
  Changes in self-reported diagnoses between baseline survey and 6- and 12 months post baseline survey. The respondent is asked whether he/she thinks they have Covid-19 sequelae, myalgic encephalomyelitis/chronic fatigue syndrome, whiplash, fibromyalgia, hypermobility, irritable bowel syndrome or food intolerance, or whether they have been diagnosed with either of these by health personnel.

OTHER OUTCOMES:
Preventive effect of sickness absence | 12 months post baseline survey
  Changes in self-reported beliefs about the potential preventive effect of short-term sickness absence on long term sickness absencebetween baseline survey and 6- and 12 months post baseline survey. The respondent is asked whether he/she agrees to 5 different statements on this topic, using a 5-point likert scale.
Health care utilization | At 12 and 60 months post first appointment at NSAC
  Based on registry data from publicly funded specialist health services and primary care, we will examine if there is any effect of the intervention on use of other health services during follow-up.
Health economic evaluation: self report EQ-5D | 12 months post baseline survey
  Health economic evaluation is measured using the EQ-5D instrument, issued to patients prior to first treatment and 6- and 12 months post baseline survey to assess change.
Health economic evaluation: self report ReQol | 12 months post baseline survey
  Health economic evaluation is measured using the ReQol instrument, issued to patients prior to first treatment and 6- and 12 months post baseline survey to assess change.
Health economic evaluation: labour costs | Time Frame: 12 months post baseline survey
  Health economic evaluation also involves data on number of professions seeing the patient and number of working hours spent on the patient by each profession seeing the patient during the treatment period, recorded in questionnaires filled out by the clinicians after each consultation. This enables calculation of costs in terms of manpower and staff.
Expectations to- and evaluation of treatment | 12 months post baseline survey
  Using open-ended questions, patients are asked about their expectations towards treatment prior to first treatment, and about their evaluation of treatment 6- and 12 months after baseline survey. These two will be compared.
Barriers for return to work | 12 months post baseline survey
  Changes in self-reported barriers for return to work between prior to first treatment and 6- and 12 months post baseline survey. The questionnaire includes 26 items concerning barriers for return to work.
Motivation for work | 12 months post baseline survey
  Changes in self-reported motivation for work between baseline survey and 6- and 12 months post baseline survey. The questionnaire consists of a number of questions concerning motivation.
Effort/reward imbalance | 12 months post baseline survey
  Changes in self-reported effort/reward imbalance (ERI) between baseline survey and 6- and 12 months post baseline survey. ERI is measured using the 3 items with the highest factor loading in the Siegrist Effort/Reward Imbalance Questionnaire (short version). A high score on either of the three items triggers the rest of the questionnaire.
Workplace bullying | 12 months post baseline survey
  Changes in self-reported workplace bullying between baseline survey and 6- and 12 months post baseline survey. Workplace bullying is measured using the Short Negative Acts Questionnaire (SNAQ).
Economic situation | 12 months post baseline survey
  Changes in self-reported economic situation between baseline survey and 6- and 12 months post baseline survey. The questionnaire includes 2 items concerning economic problems and concerns about economic problems.
Procedural justice | 12 months post baseline survey
  Changes in self-reported procedural justice between baseline survey and 6- and 12 months post baseline survey. It is measured by 3 items concerning workplace decisions.
Relational justice | 12 months post baseline survey
  Changes in self-reported relational justice between baseline survey and 6- and 12 months post baseline survey. Relational justice is measured by 4 items concerning the general behaviour of the respondent's supervisor.
Job phobia | 12 months post baseline survey
  Changes in self-reported job phobias between baseline survey and 6- and 12 months post baseline survey. Job phobia is measured by 12 items concerning the respondent's avoidance of the workplace or work-related anxiety.
Ergonomic work environment | 12 months post baseline survey
  Changes in self-reported ergonomic work environment between baseline survey and 6- and 12 months post baseline survey. Ergonomic work environment is measured by 11 items concerning the respondent's physical tasks at work.
Organisational change | 12 months post baseline survey
  Changes in self-reported organisational change between baseline survey and 6- and 12 months post baseline survey. Organisational change is measured using the 3 items covering changes in management, colleagues and tasks.
Work/family conflict | 12 months post baseline survey
  Changes in self-reported work/family conflict between baseline survey and 6- and 12 months post baseline survey. Work/family conflict is measured using the 4 items with the highest factor loading in the Home-Work Interference Scale.
Demand and control | 12 months post baseline survey
  Changes in self-reported demand and control between baseline survey and 6- and 12 months post baseline survey. Demand and control is measured using three questions from the instrument developed by Karasek/Theorell. A high score on either of the three items triggers the rest of the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Arnstein Mykletun, PhD, Principal Investigator — UiT The Arctic University of Norway
Locations (5):
- Norway (5):
  - Helse I Arbeid Nordlandssykehuset, Bodø, Nordland
  - Helse I Arbeid Helgelandssykehuset, Sandnessjøen, Nordland
  - Helsepartner Rehabilitering Alta, Alta, Troms Og Finnmark
  - Helse I Arbeid Finnmarkssykehuset, Kirkenes, Troms Og Finnmark
  - Helse I Arbeid Universitetssykehuset Nord-Norge, Tromsø, Troms Og Finnmark

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual patient data with other researchers. At the stage of analyses, associated researchers will be provided with an anonymized data set including all relevant data to answer the research questions.